CLINICAL TRIAL: NCT06459115
Title: Adherence to Medication in Patients With Acute Decompensated Heart Failure: a Cross-sectional Study at the Emergency Department (ADHF-ED= Adherence to Medication in Patients With Acute Decompensated Heart Failure at the Emergency Department)
Brief Title: Adherence to Medication in Patients With Acute Decompensated Heart Failure
Acronym: ADHF-ED
Status: Recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: ADHF-ED
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute Decompensated Heart Failure; Adherence; Emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Every day, patients present to emergency department due to acute heart failure. There are many causes for decompensation. One possible cause is a lack of adherence to heart failure medication (prognosis-improving medications and diuretics). The aim of this study is to directly measure adherence in patients with acute heart failure (gold standard of adherence measurement using liquid chromatography coupled to high-resolution mass spectrometry= LC-HRMS/MS) at the emergency department. Questionnaires are used to investigate possible factors influencing adherence.

DETAILED DESCRIPTION:
Several drugs has been shown to improve survival and to reduce the risk for hospitalization for acute heart failure (AHF) in patients with chronic heart failure.

Despite optimal drug treatment, patients with heart failure suffer one hospitalization for AHF every year on average with the requirement of intravenous diuretics. Hence, AHF is one of the leading causes for emergency department visits in elderly patients.

A possible cause for AHF in patients with known heart failure is nonadherence to drug treatment. Long-term-adherence to drugs of chronic diseases is low. Direct methods to assess adherence like the measurement drug levels or metabolites in body fluids are considered as the gold standard.

This study aimed to i) provide (direct measured) adherence rates of patients presented with AHF to the emergency department and ii) to identify patient-related factors with impact on adherence.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years of age
* known chronic heart failure irrespective of ejection fraction (heart failure with reduced, mildly reduced, or preserved ejection fraction)
* requirement of intravenous diuretics (outpatient or stationary treatment)
* stable heart failure medication >2 weeks
* ≥1 sign of volume overload (peripheral edema, jugular venous distension, pulmonary rales, ascites, or demonstration of pulmonary venous congestion on chest X-ray)
* elevated natriuretic peptides (N-terminal pro brain natriuretic peptide= nt-pro-BNP ≥125 pg/ml)

Exclusion Criteria:

- Not able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute decompensated heart failure (AHF) at the emergency department at Saarland University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to heart failure medication | 1 day (cross-sectional)
  Directly measured adherence rates (measurement of drug levels or metabolites in body fluids via toxicological analysis) of patients with acute heart failure at the emergency department
  Two different definitions of adherence are used:
  * If all prescribed drugs/metabolites for the treatment of heart failure were detectable in urine, the patient is "adherend". If 1 or at least 2 prescribed drugs were nondetectable in urine, the patient was classified as "partially adherend" and "non-adherend", respectively.
  * A 80% threshold is used. If >80% of the prescribed heart failure drugs were detectable in urine, the patient was characterized as "adherent." Otherwise, the patient was considered to be "nonadherent."

SECONDARY OUTCOMES:
Patients-related factor with impact on adherence (anxiety and depression) | 1 day (cross-sectional)
  Measurement of anxiety and depressions via one questionnaire with two subscales (Hospital Anxiety and Depression Scale- German version= HADS-D; Two subscales HADS-A (anxiety) and HADS-D (depression), each with 7 items; this results in two total scores for the HADS-A (anxiety) and HADS-D (depression) scales with value ranges from 0 - 21; higher values indicating depression or anxiety; 0-7 unremarkable, 8-10 suspicious, >10 conspicuous)
Patients-related factors with impact on adherence (social support) | 1 day (cross-sectional)
  Measurement of social support via one questionnaire (ENRICHD Social Support Instrument German version= ESSI-D; 5 items; total score 5-25; higher values indicating better social support)
Patients-related factor with impact on adherence (dementia) | 1 day (cross-sectional)
  Measurement of dementia via one questionnaire (Demtect; Total score= 0-18; 0-8= Suspected dementia; 9-12= Mild cognitive impairment; 13-18= Cognitive powers appropriate for subject's age)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine III, Cardiology, Angiology and Intensive Care Medicine, University Hospital Saarland, Saarland University, Homburg, Germany

IPD SHARING:
Plan to Share IPD: No